CLINICAL TRIAL: NCT04575714
Title: Clinical Pathways and Patients' Attitudes in Acute Low Back Pain
Acronym: AcuteLBP
Status: Completed | Type: Observational
Sponsor: CHU de Reims (Other)
Responsible Party: Sponsor
Other Study IDs: PO19084
Record Dates: First submitted 2020-09-29; First posted 2020-10-05 (Actual); Last update posted 2020-10-05 (Actual); Status verified 2020-09

CONDITIONS: Acute Low Back Pain
Keywords: Acute low back pain; low back pain; clinical pathway
MeSH Terms: conditions — Low Back Pain | interventions — Electronic Health Records

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Acute low back pain: Adult patients with acute low back pain
  Interventions: Other: Data record

INTERVENTIONS:
Other: Data record — Data record

SUMMARY:
In France the prevalence of low back pain is 70 to 80 %. It's the leading cause of health expenditure in Europe and costs 900 million euros per year to health insurance in France. This is the second reason to consult a general practitioner. Acute low back pain is defined as low back pain lasts less than 6 weeks. It represents 60 to 70 % of low back pain but only 20% of the costs induced by low back pain in general. In fact, acute low back pain often heals spontaneously.

Risk factors for acute low back pain and risk factors for chronic low back pain have been the subject of many publications. They remain very difficult to prevent in practice because of their multiplicity. Preventing acute low back pain is part of the prevention of chronic low back pain. Patient care management of low back pain is well codified and consensual in the various international recommendations. However, their application is sometimes very disparate and bad habits on both patients and professionals persist. Advices recommended in the case of low back pain are widely disseminated but their applications are little studied. In 2017, in France, health insurance started a "back pain" prevention campaign with the objective of raising awareness of good attitudes in the event of back pain. It made an initial assessment of the different knowledges concerning spinal pain in the general population but also in the medical population with the aim of improving them. It appears that number of patients would not consult physician in this case. The many proposals of care and the diversity of medical professionals, paramedics and other stakeholders, proposing to cure low back pain form as many different clinical pathways. Use of alternative or unconventional medicines is poorly assessed. In this context, it seems relevant to evaluate patient clinical pathways and patients' attitudes.

DETAILED DESCRIPTION:
The aim of the study is to explore patient clinical pathways and patients' attitudes in acute low back pain

ELIGIBILITY:
inclusion criteria :

* men and women
* aged between 18 and 65 years old
* living in France
* to have ever had an acute low back pain
* accepting to participate in the study

exclusion criteria :

- over 65 or under 18 years old

Ages: 18 Years to 65 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients between 18 and 65 years old living in France to have ever had an acute low back pain
Sampling Method: Non-Probability Sample
Enrollment: 250 (Actual)
Dates: Start 2019-07-19 (Actual); Primary Completion 2019-11-19 (Actual); Study Completion 2019-11-19 (Actual)

PRIMARY OUTCOMES:
clinical pathways | Day 0
  First professional consulted by patients : general practitioner or specialist

SECONDARY OUTCOMES:
patients' attitude | Day 0
  patient's first attitude: stop or continue physical activity

CONTACTS AND LOCATIONS:
Locations (1):
- Damien JOLLY, Reims, France